CLINICAL TRIAL: NCT04127110
Title: Activity of Lorlatinib Based on ALK Resistance Mutations on Blood in ALK Positive NSCLC Patients Previously Treated With 2nd Generation ALK Inhibitor
Brief Title: Activity of Lorlatinib Based on ALK Resistance Mutations Detected on Blood in ALK Positive NSCLC Patients
Acronym: ALKALINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1825; 2019-003862-41 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Anaplastic lymphoma kinase (ALK) positive non small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib is administered orally at the daily dose of 100 mg (four tablets of 25 mg).
  Lorlatinib will be taken continuously on a daily basis until disease progression, unacceptable toxicity, occurrence of any withdrawal criterion, whichever comes first.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib is administered orally at the daily dose of 100 mg (four tablets of 25 mg).

SUMMARY:
This study includes patients diagnosed with a metastatic non small cell lung cancer (NSCLC) with anaplastic lymphoma kinase (ALK) translocation. The standard treatment for patients with metastatic non small cell lung cancer with ALK translocation is represented by personalized treatment with drugs called ALK inhibitors. During the treatment with an ALK inhibitor, the tumour can start to grow again, because the tumour adapts to the drug and develops escape mechanisms, becoming resistant. At the tumour cells level, the mechanisms underlying resistance can include the development of other alterations, mainly mutations, including in the ALK gene. The alterations that developed depend on the drug the tumour has been exposed to.

The alterations can be identified by analysing tumour tissue obtained through a biopsy, however, repeating a tumour biopsy is difficult and risky and might not be able to provide sufficient tissue for the test. Therefore in the last years, new tests have been developed to identify the mutations in the blood.

Lorlatinib is a drug that inhibits ALK and has already been identified to be able to control the tumour growth when ALK mutations are identified and is already approved as standard treatment after progression to a previous treatment with ALK inhibitors.

The purpose of this study is to identify which patient populations may benefit most from treatment with lorlatinib, based on the alterations found in their genes.

ELIGIBILITY:
A) Enrolment in optional prospective sub-study.

The patient could be enrolled during the ongoing response to second-generation anaplastic lymphoma kinase (ALK) inhibitor if the following conditions are fulfilled:

* The patient has received at least 6 months of second generation anaplastic lymphoma kinase - tyrosine kinase inhibitor (ALK-TKI) therapy (if crizotinib-pretreated) OR
* The patient has received at least 12 months of second generation ALK-TKI therapy (if crizotinib-naïve)
* Patient is willing and able to comply with the protocol for the duration of the study including scheduled visits and examinations including follow up
* Before patient registration, written informed consent must be given according to the International Conference on Harmonisation-Good Clinical Practice (ICH/GCP), and national/local regulations

B) Enrolment in ALKALINE phase II study.

Inclusion criteria

* Age ≥18 years old
* Histologically or cytologically confirmed diagnosis of NSCLC with ALK rearrangement, assessed by fluorescence in situ hybridization (FISH) assay (Abbott Molecular Inc) or by Immunohistochemistry (IHC) (Ventana Inc) approved by food and drug administration (FDA)
* Stage IIIB (not eligible for local therapy) or stage IV (according to Union for International Cancer Control (UICC) tumor lymph node metastasis (TNM) staging v8.0)
* World health organization (WHO) performance status (WHO PS) of 0-2
* Previous treatment with at least one 2nd-generation ALK inhibitor. The 2nd-generation ALK TKI (ceritinib, alectinib, brigatinib) should be the latest therapy.
* Progressive disease during treatment with 2nd-generation ALK inhibitor prior to the administration of lorlatinib
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 by computed tomography (CT) or magnetic resonance imaging (MRI) of Chest/Abdomen/Pelvis and brain MRI performed within 28 days prior to study enrolment

  * Note: At least one measurable extracranial lesion is required.
* Archival tissue from primary tumour or metastatic site, if available, and blood samples

  * Note: if blood samples cannot be collected (patient's refusal or any other reason), patient will not be eligible for this study.
* Treated and/or untreated brain or leptomeningeal metastases will be allowed if asymptomatic and/or controlled (stable dose of steroids 7 days before the beginning of lorlatinib treatment)
* Adequate bone marrow and organ function defined as following:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10E9/L;
  * Platelets ≥ 100 x 10E9/L;
  * Hemoglobin ≥ 9 g/dL;
  * Serum total amylase ≤1.5 Upper Limit Normal (ULN);
  * Serum lipase ≤1.5 ULN;
  * Serum creatinine ≤1.5 x ULN or estimated creatinine clearance > 30 mL/min - Total serum bilirubin ≤1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN; for patients with Gilbert's disease total bilirubin may be > 1.5 x ULN, however direct bilirubin must be normal;
  * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN (≤5.0 x ULN if there is liver metastases involvement);
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 3 days prior to the first dose of lorlatinib.

  * Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression or other reasons.
* Patients of childbearing / reproductive potential should use highly effective birth control measures, as defined by the investigator, during the study treatment period and for at least 5 weeks after the last dose of lorlatinib for female patients and for at least 14 weeks after the last dose of lorlatinib for male patients. A highly effective method of birth control is defined as a method, which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:

  * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
  * Note: Lorlatinib can induce Cytochrome P450 3A4/5 (CYP3A4/5) both in vitro and in vivo. Most hormonal contraceptives are CYP3A substrates, therefore, if this method of contraception is chosen it must be used along with condom (male or female condom) due to the risk of contraception failure.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 7 days after the last dose of lorlatinib.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion criteria

* Spinal cord compression. Patients who received adequate treatment (surgery or radiotherapy) and has adequate control of the pain and stabilization and/or recovery of neurological symptoms/function for the 3 weeks prior to study entry are allowed
* Major surgery within 4 weeks prior to study enrolment. Complete wound healing from major surgery must have occurred 3 weeks before the first dose of study treatment.
* Minor surgical procedures (including port insertion, uncomplicated tooth extractions) without complete wound healing at the latest 1 week before the first dose of study treatment.
* Radiation therapy within 2 weeks of study entry. Exception are:

  * Palliative radiation (≤10 fractions) is allowed if completed at least 48 hours prior to study enrolment
  * Stereotactic or small field brain irradiation is allowed if completed at least 2 weeks prior to study enrolment
  * Whole brain radiation is allowed if completed at least 4 weeks prior to study enrolment
* Any systemic anti-cancer therapy or an investigational drug treatment completed within 5 half-lives prior to start lorlatinib (in case of clinically meaningful risk of tumour flare according to investigator's assessment, discussion with EORTC is required before enrolment)
* Any unresolved toxicities from prior systemic therapy, including haematological toxicities, greater than International Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade 2 at the time of study enrolment
* Active infection requiring therapy
* Known active hepatitis B (HBV) or hepatitis C (HCV). Active HBV is defined as a known positive hepatitis B surface antigen (HBsAg) result. Active HCV is defined by a known positive Hep C antibody (Ab) result and known quantitative HCV ribonucleic acid (RNA) result greater than the lower limits of detection of the assay
* Known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness Note: Testing for HIV must be performed at sites where mandated locally
* Any of the following cardiac criteria:

  * Clinically significant cardiovascular disease (that is active or occurred <3 months prior to enrolment): cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree atrioventricular (AV) block (unless paced) or any AV block with PR >220 msec
  * Ongoing cardiac dysrhythmias of National Cancer Institute (NCI) CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.)
  * Abnormal Left Ventricular Ejection Fraction (LVEF): LVEF <50% (assessed by multigated acquisition (MUGA) scan or echocardiogram (ECHO))
* History of interstitial lung disease (ILD) or history of (non-infectious) pneumonitis that required oral or intravenous (IV) steroids (other than Chronic obstructive pulmonary disease (COPD) exacerbation) or current pneumonitis or current evidence of interstitial lung disease. Patients with history of prior radiation pneumonitis are not excluded
* Any serious or uncontrolled acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behaviour, chronic alcoholism, drug addiction, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient not eligible for this study
* Hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption
* Inability to swallow and/or retain oral tablets or impaired gastrointestinal function or disease that may significantly alter the absorption of lorlatinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* Evidence of active hematologic or primary solid tumour malignancy (other than completely resected non-melanoma skin cancer, successfully treated in situ carcinoma for example in situ cervical cancer, completely resected and successfully treated papillary thyroid cancer, or localized and presumed cured prostate cancer) within the last 3 years
* History of hypersensitivity to excipients of Lorlatinib (please refer to Summary of Product Characteristics - SmPC)
* Patients currently receiving (or unable to stop use at least 3 plasma half-lives of the strong CYP3A4/5 inducer before lorlatinib treatment is started) medications or herbal supplements known ti be strong inducers of the cytochrome P450 (CYP) 3A4/5
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Important note: All eligibility criteria must be adhered to, in case of deviation a discussion with Headquarters and study coordinator is mandatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 months after enrolment of last patient
  Progression Free Survival Rate at 12 months (PFSR-12) is defined as the proportion of patients at 12 months who are alive and non-progressing.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months after enrolment of last patient
  OS is defined as the time interval between the date of enrolment and the date of death from any cause. If no event has been observed, then the patient is censored at the last date known to be alive.
Overall Response Rate (ORR) | 12 months after enrolment of last patient
  Overall Response Rate (ORR) is an overall rate including patients with documented complete response (CR) or partial response (PR)
Duration of Response (DOR) | 12 months after enrolment of last patient
  Duration of Response will only be reported for patients who achieved either CR or PR. The duration of response is measured from the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. If progression has not been observed, the patient will be censored at the date of the last follow up examination. In the event of death without progression competing risk method will be used.
CNS Overall Response Rate (CNS-ORR) | 12 months after enrolment of last patient
  CNS Overall Response Rate (CNS ORR) is an overall rate including patients with documented complete response (CNS-CR) or partial response (CNS-PR)
Safety profile according to NCI CTCAE v.5 | 30 days after last dose
  Safety profile according to NCI CTCAE v.5

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Dingemans, MD, Principal Investigator — Erasmus MC, Rotterdam, Netherlands; Laura Mezquita, MD, Principal Investigator — Hospital Clinic Universitari de Barcelona, Spain
Locations (26):
- Belgium (4):
  - Institut Jules Bordet-Hopital Universitaire ULB, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU-UCL Namur - CHU Mont Godinne - UCL Namur, Yvoir
- France (5):
  - Centre Hospitalier Avignon, Avignon
  - Assistance Publique Hopitaux Paris - Hopital Avicenne, Bobigny
  - CHU de Brest, Brest
  - Centre Hopitalier Intercommunal De Creteil, Créteil
  - Gustave Roussy, Villejuif
- King Hussein Cancer Center, Amman, Jordan
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus MC, Rotterdam
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Spain (11):
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra - Clinica Universitaria De Navarra, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Clinica Universidad de Navarra - Clinica Universitaria De Navarra, Pamplona
  - University Hospital Virgen del Rocio, Seville
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No